CLINICAL TRIAL: NCT00143650
Title: Does House Dust From Water Damaged Buildings Cause Stronger Responses Among Occupants Than Dust From Buildings Without Water Damage? Can Occupants' Sensitivity be Predicted by Biomarkers?
Brief Title: SENOC-I Det Sunda Huset II - Sensitization of Occupants of Water Damaged Buildings.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government)
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FORMAS 24.2/2001-05; SENOC,APU 0103.
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2005-01

CONDITIONS: Upper Airway, Irritation Inflammation, Discomfort
Keywords: Upper airway, irritation inflammation, discomfort, house dust, damp buildings, climate chamber, humans
MeSH Terms: interventions — Dust

INTERVENTIONS:
Behavioral: House dust

SUMMARY:
The study is focussed on two main questions:

1. The importance of dampness of the building and home dust as a factor of the subjects= responses.
2. Can measures used in KLINIR predict the subjects' responses to the dust?

This study therefore was arranged to test the following hypotheses:

1. Does dust in general cause inflammatory/body perceptions through e.g. an irritation symptoms index.
2. Does the dust include effective odorants which affects an IAQ index?
3. Does dampness increase the content of organic or inorganic compounds e.g. of microbial origin that causes the dust to be more reactive? (Differences between the two types of dust)
4. Is the sensitivity of the subjects explaining the responses to exposures in a, b, or c? (Subject group and sensitivity index)

As explorative investigations biomarkers for exposures and sensitivity for practical usage are tested.

DETAILED DESCRIPTION:
The study is focussed on two main questions:

c. The importance of dampness of the building and home dust as a factor of the subjects= responses.

d. Can measures used in KLINIR predict the subjects' responses to the dust?

As explorative investigations biomarkers for exposures and sensitivity are tested for practical use.

These investigations are made during experimental exposures of subjects to dust from dry and water damaged buildings. The responses of healthy KLINIR-sensitive subjects are predicted using personal sensitivity measures.

The design is a 3x3 Latin square design (cross-over design). The subjects will be their own controls and comparisons to placebo (clean air) were made. The study was double blinded and the subjects were only informed about details on design and exposures after the experiment and only if they asked.

This design eliminated effects of any learning or training during the investigations, and also the effects of season and weekday was eliminated. The subjects were exposed with 3-4 weeks interval to eliminate carry-over of effects from one exposure session to the next.

The design was replicated three times on three different groups of subjects each including 9 subjects. Each group of nine were divided into three groups of three subjects.

ELIGIBILITY:
Inclusion Criteria:

* All in local area, nasal histamine responsive, grass allergic, from study KLINIR.

Exclusion Criteria:

* Pregnancy, house dust allergy, hyper-responding air ways, disease, disabled

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27
Dates: Start 2001-01; Study Completion 2002-09

PRIMARY OUTCOMES:
Acoustic rhinometry, general symptoms, inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Lars Mølhave,, DMSc, Ph.D., Principal Investigator — The Air Pollution Unit, Department of Environmental and Occupational Medicine, Institute of Public Health, The University of Aarhus
Locations (1):
- The Air Pollution Unit, Department of Environmental and Occupational Medicine, Institute of Public Health, The University of Aarhus, Aarhus, Denmark